CLINICAL TRIAL: NCT03922711
Title: A Double-Blind, Randomized, Three-Arm, Parallel-Group Study to Assess the Efficacy and Safety of Two Doses of Pridopidine Versus Placebo for the Treatment of Levodopa-Induced Dyskinesia in Patients With Parkinson's Disease (gLIDe)
Brief Title: A Study to Assess the Safety and Effectiveness of Pridopidine Compared to Placebo in the Treatment of Levodopa-Induced Dyskinesia in Patients With Parkinson's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID-19
Sponsor: Prilenia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PL101-LID201
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Results first posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-04

CONDITIONS: Parkinson Disease
Keywords: Levodopa; Dyskinesia
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — pridopidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pridopidine Dose 1 (Experimental): Dose 1 (oral capsule) for 12 weeks following 2 or 4 week dosage regimen titration period
  Interventions: Drug: Pridopidine; Drug: Placebo
- Pridopidine Dose 2 (Experimental): Dose 2 for (oral capsule) for 12 weeks following 2 or 4 week dosage regimen titration period
  Interventions: Drug: Pridopidine
- Placebo (Placebo Comparator): Matching placebo (oral capsule) for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pridopidine — Oral capsule
  Arms: Pridopidine Dose 1; Pridopidine Dose 2
Drug: Placebo — Oral capsule
  Arms: Placebo; Pridopidine Dose 1

SUMMARY:
This is a multicenter, randomized, three-arm, parallel-group, double-blind, placebo-controlled, study to evaluate the efficacy, safety and pharmacokinetics (PK) of pridopidine vs. placebo for the treatment of Levodopa Induced Dyskinesia (LID) in patients with Parkinson Disease.

ELIGIBILITY:
Inclusion Criteria:

* Provides signed informed consent form.
* Has clinical diagnosis of Parkinson's Disease (PD).
* Has Levodopa-induced dyskinesia (LID).
* Patient and/or study partner must demonstrate ability to keep accurate home diary of PD symptoms.
* Has stable anti-PD treatments for at least 28 days prior to start of study treatment and kept constant throughout study.
* All routine and allowed prescription/non-prescription medications and/or nutritional supplements taken regularly must be at stable dosage for at least 28 days prior to start of study treatment and maintained throughout study.

Exclusion Criteria:

* Diagnosis of atypical Parkinsonism.
* Treatment with dopamine blocking drugs.
* History of surgical intervention related to PD, such as deep brain stimulation.
* History of severe depression, psychosis or hallucinations within 6 months prior to screening; active suicidal ideation; or suicidal attempt within 5 years prior to screening.
* History of certain cancers within 5 years prior to screening.
* Significant cardiac event within 12 weeks prior to Baseline or history of certain cardiac arrhythmias.
* History of epilepsy or seizures within 5 years prior to screening.
* Females who are pregnant or breastfeeding.
* Sexually active female patients who are not surgically sterile or at least 2 years postmenopausal prior to screening, and who do not agree to utilize a highly effective hormonal method of contraception in combination with a barrier method, from screening until at least 4 weeks after completion of study treatment.
* Male patients not using highly effective contraception or not agreeing to continue highly effective contraception until at least 90 days after the completion of study treatment.
* Treatment with any investigational product within 30 days of screening or plans to participate in another clinical study assessing any investigational product during the study.

Other protocol-defined inclusion/exclusion criteria could apply.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yael Cohen, Study Director — Prilenia
Locations (33):
- United States (33):
  - Prilenia Investigational Site (Site 117), Birmingham, Alabama
  - Prilenia Investigational Site (Site 144), Phoenix, Arizona
  - Prilenia Investigational Site (Site 111), Phoenix, Arizona
  - Prilenia Investigational Site (Site 115), Scottsdale, Arizona
  - Prilenia Investigational Site (Site 106), Fountain Valley, California
  - Prilenia Investigational Site (Site 109), Irvine, California
  - Prilenia Investigational Site (Site 105), Pasadena, California
  - Prilenia Investigational Site (Stie 142), Torrance, California
  - Prilenia Investigational Site (Site 136), Aurora, Colorado
  - Prilenia Investigational Site (Site 135), Englewood, Colorado
  - Prilenia Investigational Site (Site 118), Boca Raton, Florida
  - Prilenia Investigational Site (Site 131), Maitland, Florida
  - Prilenia Investigational Site (Site 122), Sunrise, Florida
  - Prilenia Investigational Site (Site 116), Tampa, Florida
  - Prilenia Investigational Site (Site 138), Atlanta, Georgia
  - Prilenia Investigational Site (Stie 123), Augusta, Georgia
  - Prilenia Investigational Site (Site 107), Iowa City, Iowa
  - Prilenia Investigational Site (Site 102), Kansas City, Kansas
  - Prilenia Investigational Site (Site 126), Omaha, Nebraska
  - Prilenia Investigational Site (Site 141), New Brunswick, New Jersey
  - Prilenia Investigational Site (Site 128), Amherst, New York
  - Prilenia Investigational Site (Site 147), New York, New York
  - Prilenia Investigational Site (Site 101), Raleigh, North Carolina
  - Prilenia Investigational Site (Site 127), Raleigh, North Carolina
  - Prilenia Investigational Site (Site 149), Dayton, Ohio
  - Prilenia Investigational Site (Site 139), Tulsa, Oklahoma
  - Prilenia Investigational Site (Site 114), Philadelphia, Pennsylvania
  - Prilenia Investigational Site (Site 146), Willow Grove, Pennsylvania
  - Prilenia Investigational Site (Site 119), Providence, Rhode Island
  - Prilenia Investigational Site (Site 120), Houston, Texas
  - Prilenia Investigational Site (Site 121), Houston, Texas
  - Prilenia Investigational Site (Site 129), San Antonio, Texas
  - Prilenia Investigational Site (Site 103), Kirkland, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McFarthing K, Prakash N, Simuni T. CLINICAL TRIAL HIGHLIGHTS - DYSKINESIA. J Parkinsons Dis. 2019;9(3):449-465. doi: 10.3233/JPD-199002. No abstract available. PMID 31356217
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 23 patients were randomized to pridopidine 100 mg BID (n=7), pridopidine 150 mg BID (n=8), or placebo (n=8). Of these, 5 patients randomized to 150 mg BID discontinued study drug during the titration period prematurely (i.e. did not reach the maintenance dose) and were therefore analyzed in the 100 mg BID group.
  The study was terminated early due to the COVID-19 pandemic.
Groups:
- Pridopidine 100 mg BID: Titration period of 2-week (original protocol) or 4-week (Amendment 1) duration, followed by 12-week maintenance treatment at a dose of 100 mg BID.
  2-week titration: 3 days pridopidine 75 mg QD, then 4 days pridopidine 75 mg BID, then 1 week pridopidine 100 mg BID 4-week titration: 1 week pridopidine 75 mg every 48 h, then 1 week pridopidine 75 mg QD, then 1 week pridopidine 75 mg BID, then 1 week pridopidine 100 mg BID.
- Pridopidine 150 mg BID: Titration period of 2-week (original protocol) or 4-week (Amendment 1) duration, followed by 12-week maintenance treatment at a dose of 150 mg BID.
  2-week titration: 3 days pridopidine 75 mg QD, then 4 days pridopidine 75 mg BID, then 1 week pridopidine 100 mg BID 4-week titration: 1 week pridopidine 75 mg every 48 h, then 1 week pridopidine 75 mg QD, then 1 week pridopidine 75 mg BID, then 1 week pridopidine 100 mg BID.
- Placebo: Titration period of 2-week (original protocol) or 4-week (Amendment 1) duration, followed by 12-week maintenance treatment, using pridopidine-matching placebo.
Period: Overall Study
Arm/Group | Pridopidine 100 mg BID | Pridopidine 150 mg BID | Placebo
Started | 7 | 8 | 8
Treatment Group Based on Maximal Possible Highest Dose Received (Used for Analysis) (A total of 8 patients were randomized to pridopidine 150 mg BID. Of these, 5 patients discontinued study drug during titration, i.e. did not reach the full maintenance dose. Therefore, they were analyzed under the 100 mg BID group. The 100 mg BID group included patients who received any dose between 75 mg QD and 100 mg BID.) | 12 | 3 | 8
Completed | 3 | 3 | 4
Not Completed | 4 | 5 | 4
Not completed — Adverse Event | 3 | 2 | 2
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 1
Not completed — Not further specified | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: A total of 8 patients were randomized to pridopidine 150 mg BID. Of these, 5 patients discontinued study drug during titration, i.e. did not reach the full maintenance dose. Therefore, they were analyzed under the 100 mg BID group. The 100 mg BID group included patients who received any dose between 75 mg QD and 100 mg BID.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pridopidine 100 mg BID | Pridopidine 150 mg BID | Placebo | Total
Number analyzed (Participants) | 12 | 3 | 8 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (7.5) | 61.3 (12.7) | 64.0 (9.7) | 66.3 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 5 | 13
  Male | 5 | 2 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 11 | 3 | 5 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 3 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Levodopa-induced Dyskinesia as Measured by UDysRS Score
Description: Mean change from baseline (BL) in the sum of Parts 1, 3 and 4 of the Unified Dyskinesia Rating Scale (UdysRS), in the ON state.
  The UDysRS comprises 2 primary sections i.e. Historical [Part 1 (ON-Dyskinesia) and Part 2 (OFF-Dystonia)] and Objective [Part 3 (Impairment) and Part 4 (Disability)] assessment. ON-Dyskinesia are choreic and dystonic movements that occur when the Parkinson's disease (PD) medicine is working. Lower UDysRS values mean better patient outcome i.e. less dyskinesia.
  The UDysRS score for this study is calculated as sum of the parts, with scores of 0-44 for Part 1, 0-28 for Part 3 and 0-16 for Part 4.
Time Frame: Baseline; Visit 7 (at Week 16) planned. Since the study was terminated early due to the COVID-19 pandemic, analysis of the primary endpoint was done at Visit 5 (Week 8/10) in those patients who were on study drug at this visit.
Population: The primary endpoint was analyzed for the population of patients randomized and on study drug at Visit 5 (Week 8/10). Of the 3 pridopidine patients included, 1 and 2 patients, respectively, received pridopidine 100 and 150 mg. Analysis of these data, separately for each pridopidine dose, is not meaningful or conclusive.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pridopidine Total: All patients on treatment with pridopidine at the time of Visit 5 (Week 8/10) regardless of the pridopidine dose.
- Placebo: All patients on treatment with pridopidine-matching placebo at the time of Visit 5 (Week 8/10).
Arm/Group | Pridopidine Total | Placebo
Number analyzed (Participants) | 3 | 7
score on a scale
  Baseline | 32.0 (10.44) | 35.9 (6.44)
  Visit 5 | 14.7 (5.13) | 26.1 (11.02)
  Change from baseline at Visit 5 | -17.3 (6.03) | -9.7 (9.43)

ADVERSE EVENTS:
Time Frame: From screening onwards, through to Week 18 (planned); this included 2 weeks' safety follow-up after treatment completion. The study was discontinued early due to the COVID-19 pandemic. Actual exposure (mean treatment duration) was 38 days in all patients receiving pridopidine and 93 days in all patients receiving placebo.
Description: A total of 8 patients were randomized to pridopidine 150 mg BID. Of these, 5 patients discontinued study drug during titration, i.e. did not reach the full maintenance dose. Therefore, they were analyzed under the 100 mg BID group. The 100 mg BID group included patients who received any dose between 75 mg QD and 100 mg BID.
Arm/Group | Pridopidine 100 mg BID | Pridopidine 150 mg BID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/3 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/3 | 1/8
Other Adverse Events (participants affected / at risk) | 10/12 | 3/3 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pridopidine 100 mg BID (N=12) | Pridopidine 150 mg BID (N=3) | Placebo (N=8)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pridopidine 100 mg BID (N=12) | Pridopidine 150 mg BID (N=3) | Placebo (N=8)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Drug ineffective (General disorders) | 1 (1) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0)
Feeling jittery (General disorders) | 1 (16) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Temperature intolerance (General disorders) | 0 (0) | 1 (2) | 0 (0)
Drug effect decreased (General disorders) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bacterial test positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (6) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (8) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anosmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Freezing phenomenon (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Initial insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal odour (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early due to the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data and results are owned by the sponsor. Results can be used by the institution for (a) internal noncommercial research, education and patient care, and (b) as required under applicable laws and regulations. Other uses require prior written consent of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2019-11-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT03922711/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT03922711/SAP_001.pdf